CLINICAL TRIAL: NCT01706198
Title: A 12-month, Open Label, Randomised, Effectiveness Study to Evaluate Fluticasone Furoate (FF, GW685698)/Vilanterol (VI, GW642444) Inhalation Powder Delivered Once Daily Via a Novel Dry Powder Inhaler Compared With Usual Maintenance Therapy in Subjects With Asthma
Brief Title: An Effectiveness Study Comparing Fluticasone Furoate (FF, GW685698)/Vilanterol (VI, GW642444) With Standard Treatment in Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 115150
Record Dates: First submitted 2012-10-04; First posted 2012-10-15 (Estimated); Results first posted 2019-01-24 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2018-07

CONDITIONS: Asthma
Keywords: respiratory; adult; asthma
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate; vilanterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FF/VI (Experimental): fluticasone furoate (FF) + vilanterol (VI) once daily via a Novel Dry Powder Inhaler
  Interventions: Drug: fluticasone furoate + vilanterol; Drug: inhaled corticosteroid with or without a long acting beta2-agonist
- ICS or ICS/LABA maintenance therapy (Active Comparator): inhaled corticosteroid (ICS) alone or in combination with a long acting beta2-agonist (LABA)
  Interventions: Drug: inhaled corticosteroid with or without a long acting beta2-agonist

INTERVENTIONS:
Drug: fluticasone furoate + vilanterol — once daily via a Novel Dry Powder Inhaler
  Arms: FF/VI
Drug: inhaled corticosteroid with or without a long acting beta2-agonist — ICS alone or in combination with a long acting bronchodilator

SUMMARY:
This study is designed to compare the effectiveness and safety of Fluticasone Furoate/Vilanterol Inhalation Powder (100mcg Fluticasone Furoate ((FF), GW685698)/25mcg Vilanterol ((VI), GW642444) or 200mcg Fluticasone Furoate ((FF), GW685698)/25mcg Vilanterol ((VI), GW642444) ) delivered once daily via a Novel Dry Powder Inhaler (NDPI) compared with the existing asthma maintenance therapy over twelve months in subjects diagnosed with asthma. This is a Phase III multi-centre, randomised open label study. Subjects who meet the eligibility criteria are randomised and will enter a 12 month treatment period.

DETAILED DESCRIPTION:
This is a Phase III multi-centre, randomised open label study performed in subjects followed in primary care who have a diagnosis of and receive regular treatment for asthma in a localised geographical region of the UK

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for enrolment in the study must meet all of the following criteria:

1. Informed consent: Subjects must be able to provide informed consent, have their consent signed and dated.
2. Type of subject: Subjects with documented GP diagnosis of asthma as their primary respiratory disease.
3. Current Anti-Asthma Therapy: All subjects must be prescribed maintenance therapy and receiving ICS with or without LABA (either a fixed combination or via separate inhalers), and for at least 4 weeks prior to Visit 2.

   * Other background asthma medication such as anti-leukotrienes are permitted
4. All subjects on ICS monotherapy or ICS/LABA combination (this can be a fixed dose combination or an ICS alone or LABA alone in separate inhalers) must have had symptoms in the past week prior to Visit 2. Symptoms are defined by daytime symptoms more than twice per week, use of short-acting beta2-agonist bronchodilator more than twice per week, any limitation of activities, or any nocturnal symptoms/awakening. (The symptoms are based on subject's recall and are consistent with the GINA and in principal with the BTS/SIGN guidelines).
5. Subject questionnaires: Subjects must be able to complete the electronic subject questionnaires as well as those questionnaires that are completed by phone or provide a proxy e.g. a partner/relative/a friend who can do so on their behalf
6. Gender and Age: Male or female subjects aged ≥18 years of age at Visit 1. A female is eligible to enter and participate in the study if she is of:

   * Non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile). Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Post-menopausal females are defined as being amenorrhoeic for greater than 1 year with an appropriate clinical profile, e.g. age appropriate, history of vasomotor symptoms. However in questionable cases, a blood sample with FSH > 40MIU/ml and estradiol <40pg/ml (<147 pmol/L) is confirmatory.

OR Child bearing potential has a negative urine pregnancy test at Visit 2, and agrees to one of the highly effective and acceptable contraceptive methods used consistently and correctly (i.e. in accordance with the approved product label and the instructions of the physician for the duration of the study - Visit 2 to the end of the study).

Exclusion Criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

1. Recent history of Life-threatening asthma: Defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest or hypoxic seizures within the last 6 months.
2. COPD Respiratory Disease: A subject must not have current evidence or GP diagnosis of chronic obstructive pulmonary disease.
3. Other diseases/abnormalities: Subjects with historical or current evidence of uncontrolled or clinically significant disease. Significant is defined as any disease that, in the opinion of the GP/ Investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
4. Drug/food allergy: Subjects with a history of hypersensitivity to any of the study medications (e.g., beta2-agonists, corticosteroid) or components of the inhalation powder (e.g., lactose, magnesium stearate). In addition, subjects with a history of severe milk protein allergy that, in the opinion of the GP/ Investigator, contraindicates the subject's participation will also be excluded.
5. Investigational Medications: A subject must not have used any investigational drug within 30 days prior to Visit 2 or within five half-lives (t½) of the prior investigational study (whichever is longer of the two), (if unsure discuss with the medical monitor prior to screening)
6. Chronic user of systemic corticosteroids: A subject who, in the opinion of the GP/Investigator, is considered to be a chronic user of systemic corticosteroids for respiratory or other indications (if unsure discuss with the medical monitor prior to screening)
7. Subjects who are using LABA without an ICS as asthma maintenance therapy.
8. Subjects who plan to move away from the geographical area where the study is being conducted during the study period and/or if subjects have not consented to their medical records being part of the electronic medical records database that is operational in the Salford area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4233 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (43):
- United Kingdom (43):
  - GSK Investigational Site, Altrincham, Cheshire
  - GSK Investigational Site, Bowdon, Cheshire
  - GSK Investigational Site, Cheadle, Cheshire
  - GSK Investigational Site, Cheadle Hulme, Cheshire
  - GSK Investigational Site, Edgeley, Cheshire
  - GSK Investigational Site, Gatley, Cheshire
  - GSK Investigational Site, Heald Green, Cheshire
  - GSK Investigational Site, Sale, Cheshire
  - GSK Investigational Site, Stockport, Cheshire
  - GSK Investigational Site, Timperley, Cheshire
  - GSK Investigational Site, Altrincham, Greater Manchester
  - GSK Investigational Site, Broadway, Davyhulme, Greater Manchester
  - GSK Investigational Site, Irlam, Greater Manchester
  - GSK Investigational Site, Irlam, Manchester, Greater Manchester
  - GSK Investigational Site, Manchester, Greater Manchester
  - GSK Investigational Site, Newall Green, Greater Manchester
  - GSK Investigational Site, Northenden, Greater Manchester
  - GSK Investigational Site, Northern Moor, Greater Manchester
  - GSK Investigational Site, Pendlebury, Greater Manchester
  - GSK Investigational Site, Salford, Greater Manchester
  - GSK Investigational Site, Salford, Manchester, Greater Manchester
  - GSK Investigational Site, Stretford, Greater Manchester
  - GSK Investigational Site, Timperley, Greater Manchester
  - GSK Investigational Site, Withington, Greater Manchester
  - GSK Investigational Site, Wythenshawe, Greater Manchester
  - GSK Investigational Site, Cadishead, Manchester
  - GSK Investigational Site, Cheadle
  - GSK Investigational Site, Eccles
  - GSK Investigational Site, Eccles, Manchester
  - GSK Investigational Site, Ellenbrook, Manchester
  - GSK Investigational Site, Irlam, Manchester
  - GSK Investigational Site, Irlam, Salford
  - GSK Investigational Site, Little Hulton, Manchester
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Pendlebury, Manchester
  - GSK Investigational Site, Salford
  - GSK Investigational Site, Salford, Manchester
  - GSK Investigational Site, Stockport
  - GSK Investigational Site, Swinton
  - GSK Investigational Site, Swinton, Manchester
  - GSK Investigational Site, Walkden, Manchester
  - GSK Investigational Site, Worsley, Manchester
  - GSK Investigational Site, Wythenshawe

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Woodcock A, Janson C, Rees J, Frith L, Lofdahl M, Moore A, Hedberg M, Leather D. Effects of switching from a metered dose inhaler to a dry powder inhaler on climate emissions and asthma control: post-hoc analysis. Thorax. 2022 Dec;77(12):1187-1192. doi: 10.1136/thoraxjnl-2021-218088. Epub 2022 Feb 7. PMID 35131893
- [Derived] Kosinski M, Nelsen L, Rizio AA, Lay-Flurrie J, von Maltzahn R, Jacques L, Schatz M, Stanford RH, Svedsater H. Psychometric properties of the Asthma Control Test in 2 randomized clinical trials. J Allergy Clin Immunol Pract. 2021 Jan;9(1):561-563.e1. doi: 10.1016/j.jaip.2020.07.040. Epub 2020 Aug 6. No abstract available. PMID 32771685
- [Derived] Svedsater H, Jones R, Bosanquet N, Jacques L, Lay-Flurrie J, Leather DA, Vestbo J, Collier S, Woodcock A. Patient-reported outcomes with initiation of fluticasone furoate/vilanterol versus continuing usual care in the Asthma Salford Lung Study. Respir Med. 2018 Aug;141:198-206. doi: 10.1016/j.rmed.2018.06.003. Epub 2018 Jun 6. PMID 30053967
- [Derived] Jacques L, Bakerly ND, New JP, Svedsater H, Lay-Flurrie J, Leather DA. Effectiveness of fluticasone furoate/vilanterol versus fluticasone propionate/salmeterol on asthma control in the Salford Lung Study. J Asthma. 2019 Jul;56(7):748-757. doi: 10.1080/02770903.2018.1490751. Epub 2018 Oct 16. PMID 29972089
- [Derived] Woodcock A, Vestbo J, Bakerly ND, New J, Gibson JM, McCorkindale S, Jones R, Collier S, Lay-Flurrie J, Frith L, Jacques L, Fletcher JL, Harvey C, Svedsater H, Leather D; Salford Lung Study Investigators. Effectiveness of fluticasone furoate plus vilanterol on asthma control in clinical practice: an open-label, parallel group, randomised controlled trial. Lancet. 2017 Nov 18;390(10109):2247-2255. doi: 10.1016/S0140-6736(17)32397-8. Epub 2017 Sep 10. PMID 28903864
- [Derived] Woodcock A, Bakerly ND, New JP, Gibson JM, Wu W, Vestbo J, Leather D. The Salford Lung Study protocol: a pragmatic, randomised phase III real-world effectiveness trial in asthma. BMC Pulm Med. 2015 Dec 10;15:160. doi: 10.1186/s12890-015-0150-8. PMID 26651333
- [Derived] New JP, Bakerly ND, Leather D, Woodcock A. Obtaining real-world evidence: the Salford Lung Study. Thorax. 2014 Dec;69(12):1152-4. doi: 10.1136/thoraxjnl-2014-205259. Epub 2014 Mar 6. PMID 24603195
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-center, randomized, open label study to evaluate the effectiveness of fluticasone furoate (FF)/vilanterol (VI) Inhalation Powder (FF 100 micrograms [mcg]/VI 25 mcg or FF 200 mcg/VI 25 mcg) compared with usual asthma maintenance therapy in participants with asthma in a localized geographical region of United Kingdom.
Pre-assignment Details: A total of 4725 participants were screened of which 4233 participants were randomized to either initiate with FF/VI or continue their usual asthma maintenance therapy in a ratio of 1:1. The total duration of study was approximately 12 months (52 weeks).
Groups:
- Usual Care: Participants continued their usual asthma maintenance therapy that is, inhaled corticosteroid without a long acting beta2-agonist or inhaled corticosteroid with long acting beta2-agonist combination (either as a fixed dose combination or an inhaled corticosteroid/long acting beta2-agonist provided in two separate inhalers).
- FF/VI: Participants initiated with an appropriate dose of inhaled FF/VI (100 mcg/25 mcg or 200 mcg/25 mcg per actuation) once daily via Novel Dry Powder Inhaler.
Period: Overall Study
Arm/Group | Usual Care | FF/VI
Started | 2119 | 2114
Completed | 1946 | 1920
Not Completed | 173 | 194
Not completed — Adverse Event | 12 | 15
Not completed — Protocol Violation | 7 | 5
Not completed — Other: Subject reached stopping criteria | 11 | 13
Not completed — Lost to Follow-up | 97 | 93
Not completed — Physician Decision | 23 | 37
Not completed — Withdrawal by Subject | 23 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | FF/VI | Total
Number analyzed (Participants) | 2119 | 2114 | 4233
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.7 (16.69) | 49.9 (16.05) | 49.8 (16.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1241 | 1257 | 2498
  Male | 878 | 857 | 1735
Race/Ethnicity, Customized [Number; unit: Count of Participants]
  African American/African Heritage | 25 | 40 | 65
  Asian - Central/South Asian Heritage | 35 | 46 | 81
  Asian - East Asian Heritage | 4 | 9 | 13
  Asian - Japanese Heritage | 2 | 0 | 2
  Asian - South East Asian Heritage | 9 | 18 | 27
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  White - Arabic/North African Heritage | 6 | 5 | 11
  White - White/Caucasian/European Heritage | 2002 | 1971 | 3973
  Mixed race | 33 | 23 | 56
  Unknown | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Have Either an Asthma Control Test (ACT) Total Score of >=20 or an Increase From Baseline of >=3 in ACT Total Score at Week 24.
Description: The ACT is a validated self-administered questionnaire utilizing 5 questions to assess asthma control during the past 4 weeks on a 5-point categorical scale (1 to 5). By answering all 5 questions, participants with asthma obtained an ACT score ranging between 5 and 25. Higher scores indicated better control of asthma. An ACT score of <=15 showed poorly controlled asthma; 16 to 19 showed partly controlled asthma and >=20 showed well controlled asthma. The total score was calculated as the sum of the scores from all 5 questions. The primary efficacy analysis (PEA) Population is defined as all Intent-to-Treat (ITT) participants (that is, all participants who were randomized and received at least one prescription of study medication) who have an ACT total score of <20 at Baseline (Day 0). The percentage of responders that is participants with an ACT total score >=20 or an increase from Baseline of >=3 has been presented
Time Frame: Baseline (Day 0) and Week 24
Population: PEA Population. Only participants with non-missing ACT score were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Usual Care | FF/VI
Number analyzed (Participants) | 1399 | 1373
Percentage of participants | 56 | 71
Statistical Analysis 1: Comparison: Usual Care vs FF/VI; Test type: Other; p < 0.001, Regression, Logistic — The analysis method was logistic regression adjusted for randomized treatment, asthma maintenance therapy (AMT) at Baseline per randomization stratification, Baseline ACT total score, Baseline ACT total score squared, gender and age; Adjusted Odds Ratio = 2.00, 95% CI 2-sided [1.70 to 2.34] — Adjusted odds ratio comparing FF/VI with Usual Care has been presented

2. Secondary Outcome: Percentage of Participants Who Have Either an ACT Total Score of >=20 or an Increase From Baseline of >=3 in ACT Total Score at Weeks 12, 40 and 52.
Description: The ACT is a validated self-administered questionnaire utilizing 5 questions to assess asthma control during the past 4 weeks on a 5-point categorical scale (1 to 5). By answering all 5 questions, participants with asthma obtained an ACT score ranging between 5 and 25. Higher scores indicated better control of asthma. An ACT score of <=15 showed poorly controlled asthma; 16 to 19 showed partly controlled asthma and >=20 showed well controlled asthma. The total score was calculated as the sum of the scores from all 5 questions. ITT Population comprised of all participants who were randomized and received at least one prescription of study medication. The percentage of responders that is participants with an ACT total score >=20 or an increase from Baseline of >=3 has been presented. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline (Day 0) and Weeks 12, 40 and 52
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Usual Care | FF/VI
Number analyzed (Participants) | 2119 | 2114
Percentage of participants
  Week 12, n=2032, 2009: number analyzed (Participants) | 2032 | 2009
  Week 12, n=2032, 2009 | 62 | 75
  Week 40, n=1938, 1904: number analyzed (Participants) | 1938 | 1904
  Week 40, n=1938, 1904 | 60 | 71
  Week 52, n=1922, 1896: number analyzed (Participants) | 1922 | 1896
  Week 52, n=1922, 1896 | 58 | 70
Statistical Analysis 1: Comparison: Usual Care vs FF/VI; Test type: Other; p < 0.001, Regression, Logistic — Logistic regression adjusted for randomized treatment, AMT at Baseline per randomization stratification, Baseline ACT total score, Baseline ACT total score squared, gender and age; Adjusted Odds Ratio = 1.92, 95% CI 2-sided [1.67 to 2.20] — Adjusted odds ratio comparing FF/VI with Usual Care for Week 12 has been presented
Statistical Analysis 2: Comparison: Usual Care vs FF/VI; Test type: Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Adjusted Odds Ratio = 1.66, 95% CI 2-sided [1.45 to 1.91] — Adjusted odds ratio comparing FF/VI with Usual Care for Week 40 has been presented
Statistical Analysis 3: Comparison: Usual Care vs FF/VI; Test type: Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Adjusted Odds Ratio = 1.76, 95% CI 2-sided [1.54 to 2.02] — Adjusted odds ratio comparing FF/VI with Usual Care for Week 52 has been presented

3. Secondary Outcome: Percentage of Participants With Asthma Control (ACT Total Score >=20) at Weeks 12, 24, 40 and 52.
Description: The ACT is a validated self-administered questionnaire utilizing 5 questions to assess asthma control during the past 4 weeks on a 5-point categorical scale (1 to 5). By answering all 5 questions, participants with asthma obtained an ACT score ranging between 5 and 25. Higher scores indicated better control of asthma. An ACT score of <=15 showed poorly controlled asthma; 16 to 19 showed partly controlled asthma and >=20 showed well controlled asthma. The total score was calculated as the sum of the scores from all 5 questions. The percentage of participants with an ACT total score >=20 has been presented. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Weeks 12, 24, 40 and 52
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Usual Care | FF/VI
Number analyzed (Participants) | 2119 | 2114
Percentage of participants
  Week 12, n=2032, 2009: number analyzed (Participants) | 2032 | 2009
  Week 12, n=2032, 2009 | 46 | 61
  Week 24, n=1957, 1936: number analyzed (Participants) | 1957 | 1936
  Week 24, n=1957, 1936 | 46 | 60
  Week 40, n=1938, 1904: number analyzed (Participants) | 1938 | 1904
  Week 40, n=1938, 1904 | 45 | 58
  Week 52, n=1922, 1896: number analyzed (Participants) | 1922 | 1896
  Week 52, n=1922, 1896 | 44 | 58
Statistical Analysis 1: Comparison: Usual Care vs FF/VI; Test type: Other; p < 0.001, Regression, Logistic — The analysis method was logistic regression adjusted for randomized treatment, AMT at Baseline per randomization stratification, Baseline ACT total score, gender and age; Adjusted Odds Ratio = 2.09, 95% CI 2-sided [1.82 to 2.40] — Adjusted odds ratio comparing FF/VI with Usual Care at Week 12 has been presented
Statistical Analysis 2: Comparison: Usual Care vs FF/VI; Test type: Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Adjusted Odds Ratio = 1.96, 95% CI 2-sided [1.70 to 2.25] — Adjusted odds ratio comparing FF/VI with Usual Care at Week 24 has been presented
Statistical Analysis 3: Comparison: Usual Care vs FF/VI; Test type: Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Adjusted Odds Ratio = 1.79, 95% CI 2-sided [1.56 to 2.06] — Adjusted odds ratio comparing FF/VI with Usual Care at Week 40 has been presented
Statistical Analysis 4: Comparison: Usual Care vs FF/VI; Test type: Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Adjusted Odds Ratio = 1.95, 95% CI 2-sided [1.69 to 2.24] — Adjusted odds ratio comparing FF/VI with Usual Care at Week 52 has been presented

4. Secondary Outcome: Percentage of Participants Who Have an Increase From Baseline of >=3 in ACT Total Score at Weeks 12, 24, 40 and 52.
Description: The ACT is a validated self-administered questionnaire utilizing 5 questions to assess asthma control during the past 4 weeks on a 5-point categorical scale (1 to 5). By answering all 5 questions, participants with asthma obtained an ACT score ranging between 5 and 25. Higher scores indicated better control of asthma. An ACT score of <=15 showed poorly controlled asthma; 16 to 19 showed partly controlled asthma and >=20 showed well controlled asthma. The total score was calculated as the sum of the scores from all 5 questions. The percentage of participants with an increase in ACT total score >=3 from Baseline has been presented. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline (Day 0) and Weeks 12, 24, 40 and 52
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Usual Care | FF/VI
Number analyzed (Participants) | 2119 | 2114
Percentage of participants
  Week 12, n=2032, 2009: number analyzed (Participants) | 2032 | 2009
  Week 12, n=2032, 2009 | 39 | 55
  Week 24, n=1957, 1936: number analyzed (Participants) | 1957 | 1936
  Week 24, n=1957, 1936 | 40 | 54
  Week 40, n=1938, 1904: number analyzed (Participants) | 1938 | 1904
  Week 40, n=1938, 1904 | 42 | 53
  Week 52, n=1922, 1896: number analyzed (Participants) | 1922 | 1896
  Week 52, n=1922, 1896 | 37 | 50
Statistical Analysis 1: Comparison: Usual Care vs FF/VI; Test type: Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Adjusted Odds Ratio = 2.28, 95% CI 2-sided [1.98 to 2.62] — Adjusted odds ratio comparing FF/VI with Usual Care at Week 12 has been presented
Statistical Analysis 2: Comparison: Usual Care vs FF/VI; Test type: Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Adjusted Odds Ratio = 2.09, 95% CI 2-sided [1.81 to 2.41] — Adjusted odds ratio comparing FF/VI with Usual Care at Week 24 has been presented
Statistical Analysis 3: Comparison: Usual Care vs FF/VI; Test type: Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Adjusted Odds Ratio = 1.76, 95% CI 2-sided [1.53 to 2.02] — Adjusted odds ratio comparing FF/VI with Usual Care at Week 40 has been presented
Statistical Analysis 4: Comparison: Usual Care vs FF/VI; Test type: Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Adjusted Odds Ratio = 1.91, 95% CI 2-sided [1.66 to 2.21] — Adjusted odds ratio comparing FF/VI with Usual Care at Week 52 has been presented

5. Secondary Outcome: Mean Change From Baseline in ACT Total Score at Weeks 12, 24, 40 and 52.
Description: The ACT is a validated self-administered questionnaire utilizing 5 questions to assess asthma control during the past 4 weeks on a 5-point categorical scale (1 to 5). By answering all 5 questions, participants with asthma obtained an ACT score ranging between 5 and 25. Higher scores indicated better control of asthma. An ACT score of <=15 showed poorly controlled asthma; 16 to 19 showed partly controlled asthma and >=20 showed well controlled asthma. The total score was calculated as the sum of the scores from all 5 questions. Baseline value is the value at Visit 2 (Day 0) assessment. Change from Baseline is the value at post-dose visit minus Baseline. The least square mean change in ACT scores has been presented. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline (Day 0) and Weeks 12, 24, 40 and 52
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Scores on ACT scale
Arm/Group | Usual Care | FF/VI
Number analyzed (Participants) | 2119 | 2114
Scores on ACT scale
  Week 12, n=2032, 2009: number analyzed (Participants) | 2032 | 2009
  Week 12, n=2032, 2009 | 1.77 (0.087) | 3.31 (0.087)
  Week 24, n=1957, 1936: number analyzed (Participants) | 1957 | 1936
  Week 24, n=1957, 1936 | 1.70 (0.093) | 3.20 (0.094)
  Week 40, n=1938, 1904: number analyzed (Participants) | 1938 | 1904
  Week 40, n=1938, 1904 | 1.63 (0.096) | 3.00 (0.097)
  Week 52, n=1922, 1896: number analyzed (Participants) | 1922 | 1896
  Week 52, n=1922, 1896 | 1.49 (0.094) | 2.99 (0.095)
Statistical Analysis 1: Comparison: Usual Care vs FF/VI; Test type: Other; p < 0.001, Mixed Model Repeated Measures (MMRM) — MMRM adjusted for randomized treatment, AMT at Baseline per randomization stratification, Baseline ACT total score, randomized treatment-by-Baseline ACT total score interaction, gender, age, visit and randomized treatment by visit interaction; Mean Difference (Net) = 1.54, 95% CI 2-sided [1.30 to 1.77] — Treatment difference of FF/VI versus Usual Care at Week 12 has been presented
Statistical Analysis 2: Comparison: Usual Care vs FF/VI; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Net) = 1.50, 95% CI 2-sided [1.25 to 1.76] — Treatment difference of FF/VI versus Usual Care at Week 24 has been presented
Statistical Analysis 3: Comparison: Usual Care vs FF/VI; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Net) = 1.37, 95% CI 2-sided [1.11 to 1.63] — Treatment difference of FF/VI versus Usual Care at Week 40 has been presented
Statistical Analysis 4: Comparison: Usual Care vs FF/VI; Test type: Other; p < 0.001, MMRM — [p-value comment as in outcome 5, analysis 1]; Mean Difference (Net) = 1.50, 95% CI 2-sided [1.24 to 1.76] — Treatment difference of FF/VI versus Usual Care at Week 52 has been presented

6. Secondary Outcome: Percentage of Participants in Each ACT Total Score Category (>=20, 16 to 19, <=15) at Weeks 12, 24, 40 and 52.
Description: The ACT is a validated self-administered questionnaire utilizing 5 questions to assess asthma control during the past 4 weeks on a 5-point categorical scale (1 to 5). By answering all 5 questions, participants with asthma obtained an ACT score ranging between 5 and 25. Higher scores indicated better control of asthma. An ACT score of <=15 showed poorly controlled asthma; 16 to 19 showed partly controlled asthma and >=20 showed well controlled asthma. The total score was calculated as the sum of the scores from all 5 questions. The percentage of participants under each ACT total score category that is >=20, 16 to 19 and <=15 has been presented. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Weeks 12, 24, 40 and 52
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Usual Care | FF/VI
Number analyzed (Participants) | 2119 | 2114
Percentage of participants
  >=20, Week 12, n=2032, 2009: number analyzed (Participants) | 2032 | 2009
  >=20, Week 12, n=2032, 2009 | 46 | 61
  16 to 19, Week 12, n=2032, 2009: number analyzed (Participants) | 2032 | 2009
  16 to 19, Week 12, n=2032, 2009 | 26 | 20
  <=15, Week 12, n=2032, 2009: number analyzed (Participants) | 2032 | 2009
  <=15, Week 12, n=2032, 2009 | 28 | 18
  >=20, Week 24, n=1957, 1936: number analyzed (Participants) | 1957 | 1936
  >=20, Week 24, n=1957, 1936 | 46 | 60
  16 to 19, Week 24, n=1957, 1936: number analyzed (Participants) | 1957 | 1936
  16 to 19, Week 24, n=1957, 1936 | 25 | 20
  <=15, Week 24, n=1957, 1936: number analyzed (Participants) | 1957 | 1936
  <=15, Week 24, n=1957, 1936 | 29 | 20
  >=20, Week 40, n=1938, 1904: number analyzed (Participants) | 1938 | 1904
  >=20, Week 40, n=1938, 1904 | 45 | 58
  16 to 19, Week 40, n=1938, 1904: number analyzed (Participants) | 1938 | 1904
  16 to 19, Week 40, n=1938, 1904 | 24 | 21
  <=15, Week 40, n=1938, 1904: number analyzed (Participants) | 1938 | 1904
  <=15, Week 40, n=1938, 1904 | 31 | 21
  >=20, Week 52, n=1922, 1896: number analyzed (Participants) | 1922 | 1896
  >=20, Week 52, n=1922, 1896 | 44 | 58
  16 to 19, Week 52, n=1922, 1896: number analyzed (Participants) | 1922 | 1896
  16 to 19, Week 52, n=1922, 1896 | 26 | 20
  <=15, Week 52, n=1922, 1896: number analyzed (Participants) | 1922 | 1896
  <=15, Week 52, n=1922, 1896 | 30 | 21

7. Secondary Outcome: Annual Rate of Asthma-related Secondary Care Contacts
Description: All contacts are defined as any encounter the participant may have with a doctor, nurse or other healthcare professionals working as part of the National Health Service (NHS) as identified in the electronic medical records (EMR). Contacts were defined to be asthma-related if the most prominent signs and symptoms that the participant presented were a direct result of the participant's asthma. An asthma-related secondary care contact is defined as an inpatient admission or a specialist outpatient visit or an accident and emergency (A&E) contact. A participant with an A&E contact and subsequent inpatient admission was considered to have had two healthcare contacts. The least square mean annual rate of all asthma-related secondary care contacts along with 95% confidence interval has been presented.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Contacts per participant per year
Arm/Group | Usual Care | FF/VI
Number analyzed (Participants) | 2119 | 2114
Contacts per participant per year | 0.30 [0.25 to 0.34] | 0.30 [0.26 to 0.36]
Statistical Analysis 1: Comparison: Usual Care vs FF/VI; Test type: Other; p = 0.786, Generalized Linear Model (GLM) — GLM assuming negative binomial distribution (NBD) adjusted for randomized treatment, asthma maintenance therapy at Baseline per randomization stratification, ACT total score at Baseline per randomization stratification, gender and age; Ratio = 1.03, 95% CI 2-sided [0.83 to 1.28] — Ratio comparing FF/VI with Usual Care has been presented

8. Secondary Outcome: Annual Rate of Asthma-related Primary Care Contacts
Description: All contacts are defined as any encounter the participant may have with a doctor, nurse or other healthcare professionals working as part of the NHS as identified in the EMR. Contacts were defined to be asthma-related if the most prominent signs and symptoms that the participant presented were a direct result of the participant's asthma. Asthma-related primary care contacts is defined as the sum of primary care contacts on a given calendar date with either a nurse, General Practitioner or other healthcare professional that can be considered as asthma-related as per Read codes. The least square mean annual rate of all asthma-related primary care contacts along with 95% confidence interval has been presented.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Contacts per participant per year
Arm/Group | Usual Care | FF/VI
Number analyzed (Participants) | 2119 | 2114
Contacts per participant per year | 1.42 [1.36 to 1.47] | 1.45 [1.39 to 1.51]
Statistical Analysis 1: Comparison: Usual Care vs FF/VI; Test type: Other; p = 0.461, Generalized Linear Model (GLM) — GLM assuming NBD adjusted for randomized treatment, asthma maintenance therapy at Baseline per randomization stratification, ACT total score at Baseline per randomization stratification, gender and age; Ratio = 1.02, 95% CI 2-sided [0.97 to 1.08] — Ratio comparing FF/VI with Usual Care has been presented

9. Secondary Outcome: Number of Participants With Time to First Asthma-related Primary Care Contact
Description: Asthma-related primary care contact is defined as the sum of primary care contacts on a given calendar date with either a nurse, General Practitioner or other healthcare professional that can be considered as asthma-related as per Read codes. Time to first asthma-related primary care contact was measured from the date of randomization (that is, study treatment start date) to the date of first asthma-related primary care contact, or study treatment stop date for participants who completed the study without any asthma-related primary care contacts (censored). Analyses of time to first asthma-related primary care contact was censored at Day 364. The number of participants at risk at Weeks 0, 13, 26, 39 and 52 has been presented. Kaplan Meier method of analysis was used. Study related primary care contacts (that is, contacts scheduled solely due to the participant taking part in clinical trial) were excluded from this analysis.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Usual Care | FF/VI
Number analyzed (Participants) | 2119 | 2114
Participants
  Week 0 | 2119 | 2114
  Week 13 | 1621 | 1599
  Week 26 | 1208 | 1214
  Week 39 | 907 | 932
  Week 52 | 479 | 488

10. Secondary Outcome: Annual Rate of All On-treatment Secondary Care Contacts
Description: A secondary care contact is defined as an inpatient admission or a specialist outpatient visit or an A&E contact. A participant with an A&E contact and subsequent inpatient admission was considered to have had two healthcare contacts. The inpatient admissions recorded at two hospitals on the same day, were counted as a single (inpatient admission) secondary care contact. In the situation where inpatient admission periods overlapped (example, a new inpatient admission was recorded within the dates of an existing inpatient admission period), it was counted as a single (inpatient admission) healthcare contact with start date defined as the earliest inpatient admission date for either of the overlapping admissions and end date defined as the latest discharge date for either of the overlapping admissions. The least square mean annual rate of all on-treatment secondary care contacts along with 95% confidence interval has been summarized.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Contacts per participant per year
Arm/Group | Usual Care | FF/VI
Number analyzed (Participants) | 2119 | 2114
Contacts per participant per year | 5.23 [4.91 to 5.57] | 5.17 [4.86 to 5.51]
Statistical Analysis 1: Comparison: Usual Care vs FF/VI; Test type: Other; p = 0.822, Generalized Linear Model (GLM) — [p-value comment as in outcome 8, analysis 1]; Ratio = 0.99, 95% CI 2-sided [0.91 to 1.08] — Ratio comparing FF/VI with Usual Care has been presented

11. Secondary Outcome: Annual Rate of All On-treatment Primary Care Contacts
Description: All contacts are defined as any encounter the participant may have with a doctor, nurse or other healthcare professionals working as part of the NHS as identified in the EMR. Total primary care contacts is defined as the sum of primary care contacts on a given calendar date with either a nurse, General Practitioner or other healthcare professional. The least square mean annual rate of all on-treatment primary care contacts along with 95% confidence interval has been presented.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Contacts per participant per year
Arm/Group | Usual Care | FF/VI
Number analyzed (Participants) | 2119 | 2114
Contacts per participant per year | 10.61 [10.26 to 10.98] | 11.64 [11.25 to 12.04]
Statistical Analysis 1: Comparison: Usual Care vs FF/VI; Test type: Other; p < 0.001, Generalized Linear Model (GLM) — [p-value comment as in outcome 8, analysis 1]; Ratio = 1.10, 95% CI 2-sided [1.05 to 1.15] — Ratio comparing FF/VI with Usual Care has been presented

12. Secondary Outcome: Number of Participants With Time to First Primary Care Contact
Description: Time to first primary care contact is measured from the date of randomization (that is, study treatment start date) to the date of first primary care contact, or study treatment stop date for participants who completed the study without any primary care contacts (censored). Analyses of time to first primary care contact will be censored at Day 364. The number of participants at risk at Weeks 0, 13, 26, 39 and 52 has been presented. Kaplan Meier method of analysis was used. Study related primary care contacts (that is, contacts scheduled solely due to the participant taking part in clinical trial) were excluded from this analysis.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Usual Care | FF/VI
Number analyzed (Participants) | 2119 | 2114
Participants
  Week 0 | 2119 | 2114
  Week 13 | 513 | 483
  Week 26 | 245 | 242
  Week 39 | 160 | 178
  Week 52 | 79 | 96

13. Secondary Outcome: Mean Annual Rate of Severe Asthma Exacerbations
Description: A severe asthma exacerbation is defined as deterioration of asthma requiring the use of systemic corticosteroids (tablets, suspension, or injection) or antibiotics, and inpatient hospitalization, or emergency department visit due to asthma that required systemic corticosteroids or antibiotics. Least square mean for annual rate of severe asthma exacerbation along with 95% confidence interval has been presented.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Exacerbations per participant per year
Arm/Group | Usual Care | FF/VI
Number analyzed (Participants) | 2119 | 2114
Exacerbations per participant per year | 0.41 [0.38 to 0.44] | 0.40 [0.37 to 0.43]
Statistical Analysis 1: Comparison: Usual Care vs FF/VI; Test type: Other; p = 0.697, Generalized Linear Model (GLM) — GLM assuming NBD adjusted for randomized treatment; asthma maintenance therapy and ACT total score at Baseline per randomization stratification; number of severe asthma exacerbations in previous year prior to randomization categorized; gender & age; Ratio = 0.98, 95% CI 2-sided [0.88 to 1.09] — Ratio comparing FF/VI with Usual Care has been presented

14. Secondary Outcome: Time to First Severe Asthma Exacerbation.
Description: A severe asthma exacerbation is defined as deterioration of asthma requiring the use of systemic corticosteroids (tablets, suspension, or injection) or antibiotics, and inpatient hospitalization, or emergency department visit due to asthma that required systemic corticosteroids or antibiotics. The date of a severe asthma exacerbation was defined as the exacerbation onset date. Participants who completed the study without a severe asthma exacerbation were censored. Time to first severe asthma exacerbation was measured from the date of randomization (that is, study treatment start date) to the onset date of first severe asthma exacerbation, or study treatment stop date for participants who completed the study without any severe asthma exacerbations (censored). Analyses of time to first severe asthma exacerbation was censored at Day 364. The number of participants with severe asthma exacerbation has been presented.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Usual Care | FF/VI
Number analyzed (Participants) | 2119 | 2114
Participants | 654 | 634
Statistical Analysis 1: Comparison: Usual Care vs FF/VI; Test type: Other; p = 0.504, Cox proportional hazards model — Cox proportional hazards model with randomized treatment, asthma maintenance therapy at Baseline per randomization stratification, ACT total score at Baseline per randomization stratification, gender and age as covariates; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.86 to 1.07] — A hazard ratio <1 indicated a lower risk with FF/VI compared with Usual Care

15. Secondary Outcome: Mean Number of Salbutamol Inhalers Prescribed for Each Participant Over the 12 Month Treatment Period.
Description: Salbutamol was prescribed as a rescue medication to be used as and when necessary throughout the study. The number of salbutamol inhalers used by each participant during the study was calculated based on the total number of inhalers (adjusted to an equivalence of 200 metered actuations) prescribed. Number of salbutamol inhalers prescribed during the study was derived taking the participants time on study medication into account so it corresponds to 12 months on treatment. The least square mean number of salbutamol inhalers prescribed per participant during the study has been presented. Only participants exposed to study drug for at least 30 days were included in the analysis.
Time Frame: Up to 12 months
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Mean number of inhalers per participant
Arm/Group | Usual Care | FF/VI
Number analyzed (Participants) | 2116 | 2108
Mean number of inhalers per participant | 8.0 (0.11) | 7.2 (0.11)
Statistical Analysis 1: Comparison: Usual Care vs FF/VI; Test type: Other; p < 0.001, ANCOVA — ANCOVA adjusted for randomized treatment, asthma maintenance therapy at Baseline per randomization stratification, ACT total score at Baseline per randomization stratification, gender,age & number of salbutamol inhalers in year prior to randomization; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.1 to -0.5] — Difference of FF/VI versus Usual Care has been presented

16. Secondary Outcome: Time to Modification of Initial Therapy
Description: Initial therapy is defined as the treatment that the participant was prescribed at randomization. Modification of initial therapy included any change in brand, dose or frequency of inhaler, that is, stepping up in class, dose or frequency, stepping down in class, dose or frequency, switching to another brand of inhaler, switching treatment arm or withdrawal from the study. Time to modification of initial therapy was measured from the date of randomization (that is, exposure start date) to the date of modification of initial therapy or date of treatment termination for participants who completed the study without modifiying initial therapy (censored). The number of participants with modification of initial therapy has been presented.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Usual Care | FF/VI
Number analyzed (Participants) | 2119 | 2114
Participants | 488 | 563
Statistical Analysis 1: Comparison: Usual Care vs FF/VI; Test type: Other; p < 0.001, Cox proportional hazards model — [p-value comment as in outcome 14, analysis 1]; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [1.09 to 1.38] — Hazard ratio for FF/VI versus Usual Care has been presented

17. Secondary Outcome: Percentage of Participants Who Have an Increase From Baseline of >=0.5 in Standardized Asthma Quality of Life Questionnaire [AQLQ(S)] Total Score at Week 52.
Description: The AQLQ(S) contained 32 items under the following four domains: activity limitation (11 items), symptoms (12 items), emotional function (5 items) and environmental stimuli (4 items). The response format consisted of a seven-point scale where a value of 1 indicated "total impairment" and a value of 7 indicated "no impairment". The total AQLQ(S) score is the mean of all 32 items in the questionnaire and each individual domain score was calculated as the mean of the items within that domain. Hence, the total and domain scores were each defined on a range from 1 to 7 with higher scores indicating a higher quality of life. Baseline value is the value at Day 0 assessment. Change from Baseline is post dose visit value minus Baseline. The percentage of responders that is, participants with an increase from Baseline of >=0.5 in AQLQ(S) total score has been presented. Only those participants available at the specified time point was analyzed.
Time Frame: Baseline (Day 0) and Week 52
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Usual Care | FF/VI
Number analyzed (Participants) | 1922 | 1896
Percentage of participants | 43 | 55
Statistical Analysis 1: Comparison: Usual Care vs FF/VI; Test type: Other; p < 0.001, Regression, Logistic — Logistic regression adjusted for randomized treatment, asthma maintenance therapy at Baseline per randomization stratification, ACT total score at Baseline per randomization stratification, gender, age and Baseline score; Adjusted Odds Ratio = 1.79, 95% CI 2-sided [1.55 to 2.06] — Adjusted odds ratio of FF/VI with Usual Care has been presented

18. Secondary Outcome: Percentage of Participants Who Have an Increase From Baseline of >=0.5 in AQLQ(S) Environmental Stimuli Domain Score at Week 52.
Description: The AQLQ(S) contained 32 items under the following four domains: activity limitation (11 items), symptoms (12 items), emotional function (5 items) and environmental stimuli (4 items). The response format consisted of a seven-point scale where a value of 1 indicated "total impairment" and a value of 7 indicated "no impairment". The total environmental stimuli domain score was calculated as the mean of the items within the environmental stimuli domain. Hence, the environmental stimuli domain scores were each defined on a range from 1 to 7 with higher scores indicating a higher quality of life. Baseline value is the value at Day 0 assessment. Change from Baseline is post dose visit value minus Baseline. The percentage of responders that is, participants with an increase from Baseline of >=0.5 in AQLQ(S) environmental stimuli domain score has been presented. Only those participants available at the specified time point was analyzed.
Time Frame: Baseline (Day 0) and Week 52
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Usual Care | FF/VI
Number analyzed (Participants) | 1922 | 1896
Percentage of participants | 50 | 59
Statistical Analysis 1: Comparison: Usual Care vs FF/VI; Test type: Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 17, analysis 1]; Adjusted Odds Ratio = 1.51, 95% CI 2-sided [1.31 to 1.73] — Adjusted odds ratio of FF/VI versus Usual Care has been presented

19. Secondary Outcome: Percentage of Participants With Serious Adverse Event (SAE) of Pneumonia
Description: A serious advent event (SAE) of pneumonia was defined as any SAE in the adverse event special interest (AESI) group of "pneumonia". The incidence of the SAEs of pneumonia for each treatment group is defined as the percentage of participants in that group who have experienced at least one SAE of pneumonia from start date of study treatment to the stop date of exposure + 28 days or date of study discontinuation, whichever is earliest. The percentage of participants with SAE of pneumonia has been presented.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | Usual Care | FF/VI
Number analyzed (Participants) | 2119 | 2114
Percentage of participants | 1 | 1
Statistical Analysis 1: Comparison: Usual Care vs FF/VI; Test type: Non-Inferiority — Non-inferiority is demonstrated if the upper limit of the two-sided 95% confidence interval for the incidence ratio is less than 2; Incidence ratio = 1.4, 95% CI 2-sided [0.8 to 2.7] — Incidence ratio was calculated as percentage of participants who had at least one SAE of pneumonia in the FF/VI group divided by the percentage of participants who had at least one SAE of pneumonia in the Usual Care group

20. Secondary Outcome: Time to First SAE of Pneumonia
Description: An SAE of pneumonia was defined as any SAE in the AESI group of "pneumonia". The date of an event for an SAE of pneumonia was the AE onset date. Participants who do not have an SAE of pneumonia during the first 364 days of the treatment period (start date of exposure to min [end date of exposure + 28 days, date of study discontinuation, start date of exposure + 363]) were censored. Time to first SAE of pneumonia was measured from the date of randomization (that is, study treatment start date) to the onset date of first SAE of pneumonia. The number of participants with first on-treatment SAE of pneumonia has been presented.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Usual Care | FF/VI
Number analyzed (Participants) | 2119 | 2114
Participants | 16 | 23
Statistical Analysis 1: Comparison: Usual Care vs FF/VI; Test type: Other; p = 0.255, Cox proportional hazards model — [p-value comment as in outcome 14, analysis 1]; Hazard Ratio (HR) = 1.45, 95% CI 2-sided [0.77 to 2.74] — Hazard ratio for FF/VI versus Usual Care has been presented

21. Secondary Outcome: Number of Participants With Fatal SAEs of Pneumonia
Description: All SAEs included in the AESI group of "pneumonia" were considered as an SAE of pneumonia. Fatal SAEs of pneumonia are SAEs that led to death of participants. The number of participants with fatal SAEs of pneumonia has been presented.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Usual Care | FF/VI
Number analyzed (Participants) | 2119 | 2114
Participants | 3 | 1

22. Secondary Outcome: Number of Participants With SAEs
Description: An SAE is any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; is a congenital anomaly/birth defect; important medical events which may require medical or surgical intervention for example, invasive or malignant cancers; all events of possible drug-induced liver injury with hyperbilirubinemia. The number of participants with on-treatment SAEs has been summarized.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Usual Care | FF/VI
Number analyzed (Participants) | 2119 | 2114
Participants | 284 | 284

23. Secondary Outcome: Number of Participants With Adverse Drug Reactions (ADRs)
Description: An ADR is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, for which there is a reasonable possibility that the untoward occurrence is causally related to the medicinal product. ADRs are a subset of AEs for a given medicinal product.
Time Frame: Up to Week 52
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Usual Care | FF/VI
Number analyzed (Participants) | 2119 | 2114
Participants | 109 | 326

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non- serious adverse drug reactions (ADRs) were collected from the start of study treatment and until the follow up contact (Up to Week 52).
Description: ITT Population comprised of all randomized participants who received at least one prescription of study medication
Arm/Group | Usual Care | FF/VI
All-Cause Mortality (participants affected / at risk) | 27/2119 | 15/2114
Serious Adverse Events (participants affected / at risk) | 284/2119 | 284/2114
Other Adverse Events (participants affected / at risk) | 0/2119 | 0/2114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=2119) | FF/VI (N=2114)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (2) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 4 (4)
Angina pectoris (Cardiac disorders) | 1 (1) | 5 (5)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0)
Arrhythmia (Cardiac disorders) | 3 (3) | 2 (2)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 14 (16) | 7 (7)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery thrombosis (Cardiac disorders) | 0 (0) | 1 (1)
Diastolic dysfunction (Cardiac disorders) | 2 (2) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 3 (3)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2)
Myocardial ischaemia (Cardiac disorders) | 2 (2) | 5 (5)
Myocarditis (Cardiac disorders) | 0 (0) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Branchial cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Endocardial fibroelastosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0)
Secondary hypogonadism (Endocrine disorders) | 1 (1) | 0 (0)
Angle closure glaucoma (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 4 (4) | 6 (6)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 4 (4)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 5 (5)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 5 (5) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 2 (2)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 5 (5) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 3 (3)
Haematemesis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Chest pain (General disorders) | 4 (4) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 3 (3) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Surgical failure (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 1 (2)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 3 (3)
Hepatic cirrhosis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Mycotic allergy (Immune system disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Biliary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 11 (13) | 7 (8)
Chronic hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 3 (3)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Genital herpes (Infections and infestations) | 1 (1) | 0 (0)
Genital infection (Infections and infestations) | 1 (1) | 0 (0)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 3 (3) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 2 (2)
Kidney infection (Infections and infestations) | 1 (1) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 7 (7) | 5 (5)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 2 (2)
Ophthalmic herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1)
Pilonidal cyst (Infections and infestations) | 2 (3) | 1 (1)
Pneumonia (Infections and infestations) | 13 (14) | 23 (24)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Post procedural sepsis (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 2 (2)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 3 (3) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3)
Sepsis (Infections and infestations) | 7 (7) | 3 (3)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 12 (13)
Urosepsis (Infections and infestations) | 2 (2) | 1 (1)
Viral infection (Infections and infestations) | 2 (2) | 1 (1)
Viral labyrinthitis (Infections and infestations) | 0 (0) | 1 (1)
Vulval abscess (Infections and infestations) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 2 (2) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 8 (8)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 6 (6)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 4 (5) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Intentional overdose (Injury, poisoning and procedural complications) | 5 (5) | 5 (5)
Intentional product misuse (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Pelvic fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 9 (10) | 4 (4)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull fractured base (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
International normalised ratio abnormal (Investigations) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 7 (7) | 11 (11)
Renal function test abnormal (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 13 (13) | 12 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 3 (3)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Palindromic rheumatism (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acinic cell carcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (6) | 4 (4)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Phyllodes tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Precursor B-lymphoblastic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Renal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Anosmia (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 5 (5)
Cerebrovascular disorder (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Drug withdrawal convulsions (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 2 (2) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 3 (3)
Migraine (Nervous system disorders) | 2 (2) | 5 (5)
Multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Multiple sclerosis relapse (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 2 (2) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 5 (5)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1)
Subdural hygroma (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Vascular dementia (Nervous system disorders) | 0 (0) | 1 (1)
Vertebral artery dissection (Nervous system disorders) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 3 (3)
Unwanted pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 2 (3)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0)
Antisocial personality disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Delusion (Psychiatric disorders) | 1 (1) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 4 (4)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (1)
Eating disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Hypomania (Psychiatric disorders) | 1 (1) | 0 (0)
Persistent depressive disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 2 (2)
Schizoaffective disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 2 (2) | 3 (3)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 9 (9) | 6 (6)
Chronic kidney disease (Renal and urinary disorders) | 5 (5) | 3 (3)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 2 (2)
Loin pain haematuria syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal impairment (Renal and urinary disorders) | 3 (3) | 3 (3)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 4 (4) | 2 (2)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Oedema genital (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 30 (34) | 24 (30)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary eosinophilia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 1 (1) | 1 (1)
Angiodysplasia (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 5 (6)
Essential hypertension (Vascular disorders) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Raynaud's phenomenon (Vascular disorders) | 1 (1) | 0 (0)
Superior vena cava occlusion (Vascular disorders) | 0 (0) | 1 (1)
Temporal arteritis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.